CLINICAL TRIAL: NCT01454830
Title: Phase I Double-blind Randomized Controlled Trial: Sociocultural and Cognitive Perception Intervention to Promote Positive Airway Pressure Adherence
Brief Title: Tailored Intervention to Promote Positive Airway Pressure Adherence
Acronym: SCIP-PA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); ANF (Unknown)
Responsible Party: Principal Investigator, Amy M. Sawyer, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 37007; 4R00NR011173 (NIH)
Record Dates: First submitted 2011-10-12; First posted 2011-10-19 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-09

CONDITIONS: Sleep Apnea, Obstructive; Patient Compliance
Keywords: Social support; Cognition; Adaptation, psychological; Health behavior; Patient education
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance; Health Behavior | interventions — Precision Medicine; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored (Experimental): Tailored, or individualized, intervention addressing patient education, skills training, and cognitive perceptions
  Interventions: Behavioral: Tailored
- Usual care (Active Comparator): The comparison group, usual care, includes the standard of care delivered to all newly-diagnosed OSA persons proceeding to CPAP treatment
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Tailored — Individualized on critical indicator (Self-efficacy measure in Sleep Apnea) measured at each intervention delivery period (pre-diagnosis, immediately post-diagnosis, post-CPAP titration, and during week 1 of home CPAP treatment. Intervention components include patient education, preparatory skills training, modification of inaccurate/unrealistic cognitive perceptions of risk, outcome expectations, and treatment self-efficacy
  Other Names: Individualized
  Arms: Tailored
Other: Usual care — Usual care comparison group will proceed from initial clinical evaluation for OSA, diagnosis by polysomnography, CPAP titration polysomnography, and home CPAP treatment initiation as per current standard of care
  Other Names: standard of care
  Arms: Usual care

SUMMARY:
The purpose of this study is to examine the feasibility of a tailored (i.e., individualized) intervention to promote adherence to continuous positive airway pressure therapy (CPAP) in adults with newly-diagnosed, CPAP treated, obstructive sleep apnea.

DETAILED DESCRIPTION:
Poor adherence to CPAP is a significant problem among OSA patients resulting in suboptimal health and functional outcomes. Intervention studies to promote CPAP adherence have shown relatively small effects in selected samples and were costly. The overall objective of this research is to examine the effect, feasibility, and acceptability of a tailored intervention on CPAP adherence among adults with newly-diagnosed, CPAP treated OSA. The central hypothesis is that critically timed tailored interventions that focus on sociocultural aspects and cognitive perceptions of the individual experience with OSA diagnosis and treatment will improve overall CPAP adherence rates. The pilot randomized controlled trial will examine CPAP adherence outcomes at 1wk, 1mo, and 3mo among those randomly assigned to the tailored intervention or usual (standard) care and examine specific feasibility and participant acceptability outcomes in order to design and conduct a subsequent larger randomized controlled trial testing the overall efficacy of the tailored intervention.

ELIGIBILITY:
Inclusion Criteria:

* males and females >/= 18 years of age
* newly diagnosed with apnea/hypopnea index >/= 10 events/hr
* CPAP naive
* able to read and speak English

Exclusion Criteria:

* previous diagnosis and/or treatment of OSA
* major new psychiatric diagnosis within 6 months of study enrollment
* require supplemental oxygen or bilevel positive airway pressure on CPAP titration polysomnogram
* diagnosis of co-existent sleep disorder on polysomnogram, including periodic limb movements >/= 10 events/hr with arousal, central sleep apnea with >/= 5 central events/hr, insomnia, sleep hypoventilation syndrome, or narcolepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Sawyer, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Sawyer AM, Deatrick JA, Kuna ST, Weaver TE. Differences in perceptions of the diagnosis and treatment of obstructive sleep apnea and continuous positive airway pressure therapy among adherers and nonadherers. Qual Health Res. 2010 Jul;20(7):873-92. doi: 10.1177/1049732310365502. Epub 2010 Mar 30. PMID 20354236
- [Background] Sawyer AM, Canamucio A, Moriarty H, Weaver TE, Richards KC, Kuna ST. Do cognitive perceptions influence CPAP use? Patient Educ Couns. 2011 Oct;85(1):85-91. doi: 10.1016/j.pec.2010.10.014. Epub 2010 Nov 10. PMID 21071166
- [Background] Sawyer AM, Gooneratne NS, Marcus CL, Ofer D, Richards KC, Weaver TE. A systematic review of CPAP adherence across age groups: clinical and empiric insights for developing CPAP adherence interventions. Sleep Med Rev. 2011 Dec;15(6):343-56. doi: 10.1016/j.smrv.2011.01.003. Epub 2011 Jun 8. PMID 21652236
- [Background] Weaver TE, Maislin G, Dinges DF, Younger J, Cantor C, McCloskey S, Pack AI. Self-efficacy in sleep apnea: instrument development and patient perceptions of obstructive sleep apnea risk, treatment benefit, and volition to use continuous positive airway pressure. Sleep. 2003 Sep;26(6):727-32. doi: 10.1093/sleep/26.6.727. PMID 14572127
- [Derived] Yang H, Watach A, Varrasse M, King TS, Sawyer AM. Clinical Trial Enrollment Enrichment in Resource-Constrained Research Environments: Multivariable Apnea Prediction (MAP) Index in SCIP-PA Trial. J Clin Sleep Med. 2018 Feb 15;14(2):173-181. doi: 10.5664/jcsm.6926. PMID 29246264

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 12/2011 through 1/2014 Location type: clinical sleep center
Period: Overall Study
Arm/Group | Tailored | Usual Care
Started | 61 | 57
Completed | 30 | 30
Not Completed | 31 | 27
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Post-allocation Exclude- AHI<10 | 18 | 12
Not completed — Post-allocation Exclude-refused PAP | 0 | 2
Not completed — Post-allocation Exclude-other treatment | 6 | 7
Not completed — Withdrawal - no polysomnography | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored | Usual Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (11.7) | 50.1 (10.5) | 51.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 19 | 23 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 24 | 27 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Body Mass Index, Continuous [Mean (Standard Deviation); unit: kg/m2] | 37.0 (8.1) | 39.0 (10.3) | 38.0 (9.2)
Marital Status, Categorical [Number; unit: participants]
  Married | 20 | 25 | 45
  Single | 2 | 2 | 4
  Separated or Divorced | 6 | 3 | 9
  Widow(er) | 2 | 0 | 2
Daytime Sleepiness by Epworth Sleepiness Scale, Continuous [Mean (Standard Deviation); unit: units on a scale] — Total score (sum) range is 0-24; higher scores indicate worse daytime subjective sleepiness
  units on a scale | 18.7 (5.1) | 20.4 (5.3) | 19.6 (5.2)
Apnea-hypopnea Index (AHI), events/hr, Continuous [Mean (Standard Deviation); unit: events/hour] | 33.9 (21.3) | 38.0 (28.8) | 35.9 (25.2)
Apnea-hypopnea Index (AHI), Categorical [Number; unit: participants]
  Mild: 5-15 events/hr | 3 | 8 | 11
  Moderate: >15-30 events/hr | 13 | 7 | 20
  Severe: >30 events/hr | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Nightly CPAP Use
Description: Mean CPAP use, hrs/night
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: hours/night
Arm/Group | Tailored | Usual Care
Number analyzed (Participants) | 30 | 30
hours/night | 6.4 (2.01) | 5.8 (1.35)
Statistical Analysis 1: Comparison: Tailored vs Usual Care; Pilot RCT designed to establish effect size and feasibility outcomes; no a priori power calculation; statistical significance with hypotheses testing was not objective of the pilot trial; Test type: Superiority or Other; p = 0.20, t-test, 2 sided; Mean Difference (Final Values) = 0.58, Standard Error of Mean 0.44 — unit of measurement, hours/night; positive estimation parameter favors TI group; negative estimation parameter favors UC group

2. Primary Outcome: Nightly CPAP Use
Description: Mean CPAP use, hrs/night
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: hours/night
Arm/Group | Tailored | Usual Care
Number analyzed (Participants) | 30 | 30
hours/night | 5.1 (2.05) | 5.1 (1.66)
Statistical Analysis 1: Comparison: Tailored vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.90, t-test, 2 sided; Mean Difference (Final Values) = -0.06, Standard Error of Mean 0.48 — unit of measurement: hours/night; positive estimation parameter favors TI group; negative estimation parameter favors UC group

3. Primary Outcome: Nightly CPAP Use
Description: Mean CPAP use, hrs/night
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: hours/night
Arm/Group | Tailored | Usual Care
Number analyzed (Participants) | 30 | 30
hours/night | 4.8 (2.27) | 4.7 (1.85)
Statistical Analysis 1: Comparison: Tailored vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.89, t-test, 2 sided; Mean Difference (Final Values) = 0.07, Standard Error of Mean 0.53 — units of measurement: hours/night; positive estimation parameter favors TI group; negative estimation parameter favors UC group

4. Secondary Outcome: Proportion of Sleep Time on CPAP
Description: % of Total Sleep Time (TST) using CPAP
Time Frame: 1 week
Population: Randomized participants with complete primary outcome data and secondary outcome data (total sleep time) measured by concurrent wrist actigraphy during first week of PAP treatment
Measure: Mean (Standard Deviation); unit: percentage of TST on PAP
Arm/Group | Tailored | Usual Care
Number analyzed (Participants) | 21 | 24
percentage of TST on PAP | 64.58 (12.99) | 65.73 (14.25)
Statistical Analysis 1: Comparison: Tailored vs Usual Care; Exploratory outcome of PAP use defined within the sleep period, TST (total sleep time); Test type: Superiority or Other; p = 0.78, t-test, 2 sided; Mean Difference (Final Values) = -1.15, Standard Error of Mean 4.09 — units of measurement: % TST; positive estimation parameter favors TI group; negative estimation parameter favors UC group

5. Secondary Outcome: Proportion of Participants Who Complete Protocol After Allocation
Description: Feasibility assessment - retention after enrollment and allocation employed as a feasibility outcome of pilot RCT
Time Frame: Duration of protocol period
Population: Considers only participant withdrawals, administrative withdrawals for incomplete protocol procedures due to attrition; does NOT include excluded by a priori determined exclusion criteria for protocol
Measure: Number; unit: percentage of participants
Arm/Group | Tailored | Usual Care
Number analyzed (Participants) | 61 | 57
percentage of participants | 88.5 | 86

6. Secondary Outcome: Proportion of Participants Who Withdrawal
Description: Feasibility assessment - withdrawal by participants for feasibility outcome of pilot RCT
Time Frame: Duration of protocol period
Population: Considers only participant withdrawals requested from study
Measure: Number; unit: percentage of participants
Arm/Group | Tailored | Usual Care
Number analyzed (Participants) | 61 | 57
percentage of participants | 6.56 | 7.02

7. Secondary Outcome: Acceptability of Study Intervention and Comparative Group
Description: Feasibility assessment to determine participant acceptance of the study intervention and comparative condition (i.e., usual care); semi-structured interviews conducted with 50% of participants randomly assigned to "interview" at study termination and debriefing (3 months)
Time Frame: 3 months
Population: Acceptability rating by participants allocated to "interview" at study termination and debriefing; self-reported rating for binary response to satisfaction with study experience (yes/no); reported as percentage responding "yes"; no data available for participants who withdrew or were excluded prior to 3-month visit.
Measure: Number; unit: percentage of allocated responding "yes"
Arm/Group | Tailored | Usual Care
Number analyzed (Participants) | 9 | 8
percentage of allocated responding "yes" | 100 | 100

ADVERSE EVENTS:
Time Frame: 3 months
Description: Electronic medical record review at research visit to identify serious adverse events (e.g., hospitalization, emergency department visit) Checklist adverse events at research visit to identify adverse event occurrence since last research visit
Arm/Group | Tailored | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/57
Other Adverse Events (participants affected / at risk) | 0/61 | 0/57

LIMITATIONS AND CAVEATS:
Sampling bias with convenience sampling leading to relatively few PAP users meeting definition of non-adherence (threshold definition </= 4hrs/night PAP use); Modest intervention fidelity (i.e., delivery) for telephone-delivered exposure period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No